CLINICAL TRIAL: NCT00799474
Title: Men's Beliefs About Associations Between HPV, Cancers, and HPV Vaccination
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Merck-558377
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Results first posted 2010-01-15 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2010-01

CONDITIONS: Anus Neoplasms
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This research focuses on men who have sex with men (MSM) who are at higher risk of anal cancer. The survey will evaluate their beliefs about anal and oral cancer, their knowledge about role of human papillomavirus (HPV) infection in these cancers, and their knowledge of HPV vaccination and anal Pap smears. Approximately 12% of subjects will be HIV-positive.

DETAILED DESCRIPTION:
Little research has examined men's understanding of what causes anal and oral cancers and whether HPV vaccination can play a potential protective role. This research focuses on men who have sex with men (MSM) who are at notably elevated risk of anal cancer, and seeks to characterize their beliefs about anal and oral cancer, knowledge about the etiological role of HPV infection in these cancers, as well as their knowledge of HPV vaccination and anal Pap smears. We will also study heterosexual men.

ELIGIBILITY:
Inclusion Criteria:

* male
* aged 18-59
* answered question about sexual orientation

Exclusion Criteria:

* none

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Approximately 600 men (ages 18-59) who have agreed to participate in a periodic panel through the private survey company, Knowledge Networks.
Sampling Method: Probability Sample
Enrollment: 609 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Brewer, PhD, Principal Investigator — The University of North Carolina at Chapel Hill, School of Public Health

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was collected for this cross-sectional study through an online survey. Of the 874 men invited to participate, 609 (70%) completed the online survey. A pilot test was conducted between December 29, 2008 and January 4, 2009, and the main survey was conducted between January 6, 2009 and January 26, 2009.
Groups:
- Study Participants: All study participants, this observational study was not a trial that involved multiple arms
Period: Overall Study
Arm/Group | Study Participants
Started | 609
Completed | 609
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 609
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 609
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 609
Region of Enrollment [Number; unit: participants]
  United States | 609

OUTCOME MEASURES:

1. Primary Outcome: Willingness to Receive the Human Papillomavirus (HPV) Vaccine
Description: Measured participants' willingness to receive HPV vaccine. Participants were asked how willing they would be to get HPV vaccine if it were approved for use in males. A 5-point scale ranging from "definitely not willing" to "definitely willing" was used to meausure willingness.
Time Frame: at time of interview
Population: One man reported having received human papillomavirus (HPV) vaccine so he was not asked willingness items which made the analytic sample size n=608
Measure: Number; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 608
Participants | 338

2. Secondary Outcome: Awareness of HPV Vaccine
Description: Measured if participants had heard of HPV vaccine prior to survey. Participants were asked if they had heard to HPV vaccine prior to the survey and had response options of "yes", "no", and "I don't know".
Time Frame: At time of interview
Measure: Number; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 609
Participants | 415

3. Secondary Outcome: Knowledge of HPV
Description: Assessed participants' knowledge of HPV by summing correct responses to nine HPV knowledge items. Questions addressed what diseases are associated with HPV, how HPV is transmitted, and how common HPV infection is. For each item, participants were classified as having answered the item correctly or incorrectly.
Time Frame: At time of interview
Population: HPV knowledge items were only asked to those men who had heard of HPV prior to survey (n=430)
Measure: Mean (Standard Deviation); unit: Correct Responses
Arm/Group | Study Participants
Number analyzed (Participants) | 430
Correct Responses | 4.01 (2.42)

ADVERSE EVENTS:
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 0/609
Other Adverse Events (participants affected / at risk) | 0/609

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less